CLINICAL TRIAL: NCT06383117
Title: Georgia Clinical and Translational Science Alliance (Georgia CTSA) - KL2 Scholar Award
Brief Title: Understanding Effects of Calcium on the Gut-Bone Axis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Joseph Kindler, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UL1TR002378 (NIH); KL2TR002381 (NIH)
Record Dates: First submitted 2024-04-12; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy; Adult; Calcium; Bone Resorption; Endocrine; Obesity
Keywords: calcium; post-prandial; bone; GIP; GLP-1; CTX; P1NP; PTH; mixed meal tolerance test; MMTT; glucose; Vitamin D
MeSH Terms: conditions — Bone Resorption; Obesity | interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: Randomized placebo crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, participants, team distributing pills blinded to treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo control, then calcium carbonate (Experimental): At visit 1, participants will be instructed to consume 2 capsules (containing the placebo: vegetable based cellulose) immediately before consuming a standardized meal. Within 8 weeks, at visit 2, participants will be instructed to consume 2 capsules (containing the calcium carbonate, 1200 mg total) immediately before consuming a standardized meal.
  Interventions: Dietary Supplement: Calcium carbonate; Dietary Supplement: Placebo Control
- Calcium carbonate, then placebo control (Experimental): At visit 1, participants will be instructed to consume 2 capsules (containing the calcium carbonate, 1200 mg total) immediately before consuming a standardized meal. Within 8 weeks, at visit 2, participants will be instructed to consume 2 capsules (containing the placebo: vegetable based cellulose) immediately before consuming a standardized meal.
  Interventions: Dietary Supplement: Calcium carbonate; Dietary Supplement: Placebo Control

INTERVENTIONS:
Dietary Supplement: Calcium carbonate — 2 capsules containing 600 mg of calcium carbonate each
Dietary Supplement: Placebo Control — 2 capsules containing methylcellulose

SUMMARY:
The study team is inviting 13 healthy people to complete a study to explore how calcium affects hormones and bones after eating. Participants will be asked to complete two study visits within eight weeks. Before each visit, participants will be asked to not eat or drink (except water) for 9 hours. At each visit, participants will eat the same meal provided by the research team. Along with their meal, they will take a pill - in one session, this will be a calcium supplement, and in the other, a placebo (a pill with no calcium), but they won't know which one they are taking at which session. A phlebotomist will draw blood before the meal and pill, then again several times after eating. Blood draws will take place over three hours. During that time, participants will complete questionnaires about health, diet, and physical activity.

Blood will be analyzed to check on various health indicators, like bone health markers and certain hormones, to see how they change after the meal. The difference in these health indicators between the calcium and placebo sessions will help the study team understand the impact of calcium on health after eating. This could help increase knowledge of the impact of calcium on hormones and bone health.

DETAILED DESCRIPTION:
The investigators will enroll 13 healthy adults to complete a randomized crossover trial aimed at determining effects of calcium on post-prandial changes in bone metabolism. Each subject will complete two mixed meal tolerance tests (MMTTs) on two separate days, completed within 8 weeks of one another. During both MMTTs, subjects will consume an identical test meal that has a known amount of energy, macronutrients, and micronutrients. The meal will be provided by study staff. At the start of the test meal, subjects will take either a calcium or placebo pill that is provided by the study staff. Blood measurements will be acquired at time points relative to the start of the pill/meal ingestion, which is referred to as minute 0. Blood will be collected at several time points during the 3-hour post-prandial period. Blood will be assayed for measures such as biomarkers of bone metabolism, ionized calcium, and hormones. Changes in these measures during the post-prandial period will be compared between the two meals.

Randomization: After a subject is determined to be eligible for the study and is enrolled, they will be randomized to either group A or group B. Group randomization will dictate the order in which either the calcium or placebo supplement are taken (at either visit 1 or visit 2). The subject and study team will be blinded.

Visit number 1 and 2 will use identical study protocols and procedures, with the exception of the supplement (calcium vs. Placebo) that is provided based on randomization. Questionnaires will only be completed at visit 1 with the exception of a short questionnaire capturing any possible changes in health status between the two visits. Visit 2 will be held within 8 weeks after visit 1.

MMTT: Prior to the appointment, subjects will be instructed to not consume any food or drink, other than water. They will also be reminded to not consume gum, candy, coffee etc. prior to the appointment. The test includes consuming a test meal and having blood drawn over the course of 3 hours. Following a 9-hour overnight fast, participants will be asked to have blood drawn by a qualified and experienced phlebotomist or nurse who will follow standard sterile techniques. Participants will have one fasting blood draw measurement before consuming the supplement (calcium or placebo) and meal. Following this measurement, participants will be asked to consume the test pill(s) and meal (and 12oz water), in no more than 10 minutes. In total, 75 mL of blood will be collected during each experiment. Using standard serum tubes ("red top tubes") and tubes pre-treated with protease inhibitors, blood collection will be completed at time points relative to commencement of ingestion of the meal, which will be referred to as "minute 0." Blood will be collected at minutes -1, 10, 15, 20, 30, 60, 90, 120, and 180. At minutes 10, 15, and 20, 2 mL will be collected using tubes pre-treated with protease inhibitors. At minutes -1, 30, 60, 90, 120, and 180, 7 mL will be collected using red top tubes and tubes pre-treated with protease inhibitors. After each of the blood collection time points, including time point -1, an additional 3 mL will be collected as 'waste' to clear the blood collection line for subsequent collections. Following the final measurement, participants will be offered a snack. Food cannot be consumed during the test. The participant will be monitored by trained medical staff (phlebotomists or nurses). Following completion of the study, blood specimens will be shipped to other labs that the investigators regularly collaborate with, such as University of Pennsylvania Translational Core Laboratory or UGA's Cytometry Core or Athens-Piedmont medical center.

Questionnaires: A Health History questionnaire (HHQ) will be administered to determine fracture history, medication use, menstrual health (females), etc. A demographics questionnaire will gather information on race, ethnicity, and sex. The demographic questionnaire and HHQ will be administered at the first in-person lab visit. The International Physical Activity Questionnaire will be completed for subjective assessment of physical activity and sedentary behaviors. A Food Frequency Questionnaire will be administered to assess nutrition patterns. These questionnaires will be completed by the study participants on RedCap. At visit two, a short health questionnaire will be administered to assess if there were any health changes since visit 1. In our statistical analyses, the investigators will consider data on diet, physical activity, etc. as potential confounding variables, and the investigators will use them as covariates if necessary. Mainly, these data will be used for descriptive purposes. In the instance that a change in health status between visit 1 and 2 (e.g., new medication), this information will be used to guide interpretation of results and to determine whether 'sensitivity' statistical analyses are warranted.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Aged 18-45
* Speaks/reads English

Exclusion Criteria:

* Diagnosis with a medical condition known to impact bone health, nutritional status, activity levels, or food digestion, absorption, or metabolism
* Self-reported body mass index (BMI) that is either <18.5 or >29.9
* Self-reported body weight less than 115 lbs.
* Inability to swallow pill capsules
* Less than 18 years of age
* Greater than 45 years of age
* For females, peri-menopausal or post-menopausal
* Are allergic or unwilling to consume any of the following foods: wheat, gluten, peanuts
* Inability to swallow pill capsules
* Regularly takes any daily prescription medication
* Females using any form of hormonal birth control
* Females with a non-normal or absent menstrual cycle (based on self-report)
* Females will be excluded if they are currently pregnant or breastfeeding (based on self-report)
* Females will be excluded if they gave birth to a child in the last year (based on self-report)
* People with a history of kidney stones or prior diagnosis of other kidney problems

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Difference in GIP (gastric inhibitory peptide) area under the curve between calcium and placebo | Area under the curve value during calcium arm compared to area under the curve value during placebo arm. GIP area under the curve will be computed using GIP values from minutes -1, 10, 15, 20, 30, 60, 90, 120, and 180 during a mixed-meal test.
  Comparison of GIP response to a mixed-meal test between calcium and placebo.
Difference in GLP-1 (glucagon-like peptide 1) area under the curve between calcium and placebo | Area under the curve value during calcium arm compared to area under the curve value during placebo arm. GLP-1 area under the curve will be computed using GLP-1 values from minutes -1, 10, 15, 20, 30, 60, 90, 120, and 180 during a mixed-meal test.
  Comparison of GLP-1 response to a mixed-meal test between calcium and placebo.

SECONDARY OUTCOMES:
Difference in CTX (carboxy-terminal collagen crosslinks) area under the curve between calcium and placebo | Area under the curve value during calcium arm compared to area under the curve value during placebo arm. CTX area under the curve will be computed using CTX values from minutes -1, 30, 120, 180 during a mixed-meal test.
  Comparison of CTX response to a mixed-meal test between calcium and placebo.
Difference in P1NP (N-terminal propeptide) area under the curve between calcium and placebo | Area under the curve value during calcium arm compared to area under the curve value during placebo arm. P1NP area under the curve will be computed using P1NP values from minutes -1, 30, 120, 180 during a mixed-meal test.
  Comparison of P1NP response to a mixed-meal test between calcium and placebo.

OTHER OUTCOMES:
Difference in insulin area under the curve between calcium and placebo | Area under the curve value during calcium arm compared to area under the curve value during placebo arm. Insulin area under the curve will be computed using insulin values from minutes -1, 30, 60, 90, 120, 180 during a mixed-meal test.
  Comparison of insulin response to a mixed-meal test between calcium and placebo.
Difference in glucose area under the curve between calcium and placebo | Area under the curve value during calcium arm compared to area under the curve value during placebo arm. Glucose area under the curve will be computed using glucose values from minutes -1, 30, 60, 90, 120, 180 during a mixed-meal test.
  Comparison of glucose response to a mixed-meal test between calcium and placebo.
Difference in PTH (parathyroid hormone) area under the curve between calcium and placebo | Area under the curve value during calcium arm compared to area under the curve value during placebo arm. PTH area under the curve will be computed using PTH values from minutes -1, 30, 120, 180 during a mixed-meal test.
  Comparison of PTH response to a mixed-meal test between calcium and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Kindler, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia Clinical and Translational Research Unit, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD (individual participant data) that underlie results in a publication will be made available to other researchers upon reasonable request. The team will follow Institutional policies and procedures for data sharing, including appropriate approvals and complete de-identification of data and/or specimens.
Time Frame: Data will be made available upon reasonable request by one year after the results are published
Access Criteria: Detailed request for data will be made directly to the Principal Investigator who will be responsible for reviewing and responding to requests.